CLINICAL TRIAL: NCT02964104
Title: A Multiple Dose Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC0148-0287 C (Insulin 287) for Subcutaneous Administration in Subjects With Type 2 Diabetes
Brief Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics (the Exposure of the Trial Drug in the Body) and Pharmacodynamics (the Effect of the Investigated Drug on the Body) of Insulin 287 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1436-4314; 2016-000436-18 (EudraCT Number); U1111-1178-9795 (Other: World Health Organization)
Record Dates: First submitted 2016-11-11; First posted 2016-11-15 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin icodec; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin 287 + placebo (Experimental): Each dose group will consist of 16 subjects randomised for once-weekly s.c. (subcutaneous, under the skin) administration of insulin 287 and once daily s.c. placebo (n=12) or once-weekly s.c. placebo and once daily s.c. insulin degludec (n=4)
  Interventions: Drug: Insulin icodec; Drug: placebo
- Insulin degludec + placebo (Active Comparator): Each dose group will consist of 16 subjects randomised for once-weekly s.c. (subcutaneous, under the skin) administration of insulin 287 and once daily s.c. placebo (n=12) or once-weekly s.c. placebo and once daily s.c. insulin degludec (n=4)
  Interventions: Drug: insulin degludec; Drug: placebo

INTERVENTIONS:
Drug: Insulin icodec — Administered once weekly subcutaneously (s.c., under the skin) for 35 days
  Other Names: insulin 287
  Arms: Insulin 287 + placebo
Drug: placebo — Administered once daily subcutaneously for 35 days
  Arms: Insulin 287 + placebo
Drug: insulin degludec — Administered once daily subcutaneously for 35 days
  Arms: Insulin degludec + placebo
Drug: placebo — Administered once weekly subcutaneously for 35 days
  Arms: Insulin degludec + placebo

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of insulin 287 in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age between 18 and 64 years (both inclusive) at the time of signing informed consent.
* Subject who is considered to be generally healthy (with the exception of conditions associated with diabetes mellitus), based on the medical history, physical examination, and the results of vital signs, ECG and laboratory safety tests, as judged by the investigator.
* Body mass index between 20.0 and 34.9 kg/m^2 (both inclusive).
* Type 2 diabetes mellitus (as diagnosed clinically) for ≥12 months (365 days).
* No change in insulin treatment regimen during the last 90 days prior to screening.
* Current total daily insulin treatment between 0.3 and 1.0 (I) U/kg/day (both inclusive).

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products.
* Female who is pregnant, breast-feeding, or intending to become pregnant or is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by regulation or practice)(highly effective contraceptive methods are considered those with a failure rate less than 1% undesired pregnancies per year including surgical sterilisation,hormonal intrauterine devices (coil), oral hormonal contraceptives, sexual abstinence or a surgically sterilised partner). Females who are not postmenopausal can participate in the study if they use adequate contraceptive methods. Postmenopausal is defined as women aged <52 years and being amenorrheic for more than one year with serum follicle stimulating hormone (FSH level >40 IU/L or aged ≥ 52 years and being amenorrheic for less than one year and with serum FSH level > 40 IU/L or aged ≥ 52 years being amenorrheic for more than one year.
* Receipt of any investigational medicinal product within 3 months before the screening visit of this trial.
* History of deep leg vein thrombosis or repeated episodes of deep leg vein thrombosis in 1st degree relatives (parents, siblings or children) as judged by the investigator.
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event within the past 180 days) or hypoglycaemic unawareness as judged by the investigator or hospitalisation for diabetic ketoacidosis within the past 180 days.
* Use of oral antidiabetic drugs (OADs) or GLP-1 receptor agonists (e.g. exenatide, liraglutide) within 3 months prior to screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAE) | From the first trial product administration at day 1 until completion of the post-treatment follow-up visit (day 68 - 79)

SECONDARY OUTCOMES:
AUCI287,τ,SS, area under the steady-state serum insulin 287 concentration-time curve | During one dosing interval at steady-state from 0 to 168 hours after last dose (day 29)
AUCGIR,0-24h,SS, area under the glucose infusion rate-time curve at steady state | At day 30 and day 35

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Nishimura E, Pridal L, Glendorf T, Hansen BF, Hubalek F, Kjeldsen T, Kristensen NR, Lutzen A, Lyby K, Madsen P, Pedersen TA, Ribel-Madsen R, Stidsen CE, Haahr H. Molecular and pharmacological characterization of insulin icodec: a new basal insulin analog designed for once-weekly dosing. BMJ Open Diabetes Res Care. 2021 Aug;9(1):e002301. doi: 10.1136/bmjdrc-2021-002301. PMID 34413118